CLINICAL TRIAL: NCT04813237
Title: Clinical Implications of Fetal Positioning During Delivery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Żelazna Medical Centre, LLC (Other)
Collaborators: Foundation for St. Sophia Specialist Hospital in Warsaw (Unknown)
Responsible Party: Principal Investigator, Barbara Baranowska, Assistant at Maternity Ward St. Sophia Specialst Hospital in Warsaw, Principal Investigator, Żelazna Medical Centre, LLC
Other Study IDs: PN/29/2020
Record Dates: First submitted 2021-03-12; First posted 2021-03-24 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Fetal Position and Presentation Abnormalities
Keywords: fetal malposition; fetal left occiput position; fetal right occiput position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: n a — the participants are not subjected to any type of intervention

SUMMARY:
The project aims to find a relationship between the positioning of the foetus before and during birth and the results of obstetrics and to determine their incidence in the Polish population. The study will be conducted by combining the use of ultrasound diagnostics, midwives observations during childbirth, analysis of medical documentation and a questionnaire on the activity of examined women. The obtained results will be used to prepare guidelines for the birth in a particular foetus position.

DETAILED DESCRIPTION:
The purpose of the examination is to describe the difficulties associated with delivery in a non-optimal position of the fetus. Initial observations show that such childbirth is perceived as difficult by both the women giving birth and the staff. The aim of the study is to describe the level of difficulty of this labor, expressed as the experience of the woman, as well as all the elements that may affect the difficulty of this labor, for example, slower or no progress in labor, disturbances in systolic function, injuries, the need to use epidural anesthesia, increased blood loss.

ELIGIBILITY:
Inclusion Criteria:

* during childbirth,
* in a single pregnancy,

Exclusion Criteria:

* pelvic position of the fetus
* in whom labor is induced for reasons other than post-term pregnancy,
* women who came to the hospital in the second stage of labor
* severe diseases mother or foetus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: women coming to the 3rd level hospital with a birth house. During a physiological pregnancy, with no severe coexisting diseases.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Mode of delivery | immediately after delivery
  Mode of delivery as measured by number of women who had a vaginal, instrumental or operational delivery.

SECONDARY OUTCOMES:
Duration of delivery | immediately after birth
  the time of 1,2,3 and 4 stage of labor
Uterine contractions | during birth
  uterine contractions as measured by number of contractions and assessment of uterine contractile coordination
Labor progress | during birth
  Labor progress as measured by assessment of the head insertion, advancement in the birth canal,
Epidural | immediately after delivery
  as measured by epidural or not
Perineum injury | immediately after delivery
  as measured by number and extent of injury
Episiotomy | immediately after delivery
  as measured by episiotomy or not
Methods of placental separation | immediately after delivery
  as measured by number of Duncan or SchultZ methods
Blood loss | immediately after delivery
  postpartum blood loss (ml)
Difficulty of childbirth | immediately after delivery
  difficulty of childbirth as measured by subjective assessment of the woman and the midwife

CONTACTS AND LOCATIONS:
Overall Officials: Baranowska Baranowska, PhD, Study Chair — Żelazna Medical Centre, LLC
Locations (1):
- Żelazna Medical Centre, LLC, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmad A, Webb SS, Early B, Sitch A, Khan K, Macarthur C. Association between fetal position at onset of labor and mode of delivery: a prospective cohort study. Ultrasound Obstet Gynecol. 2014 Feb;43(2):176-82. doi: 10.1002/uog.13189. PMID 23929533
- [Background] Matsuo K, Shimoya K, Ushioda N, Kimura T. Maternal positioning and fetal positioning in utero. J Obstet Gynaecol Res. 2007 Jun;33(3):279-82. doi: 10.1111/j.1447-0756.2007.00524.x. PMID 17578355
- [Background] Guittier MJ, Othenin-Girard V, de Gasquet B, Irion O, Boulvain M. Maternal positioning to correct occiput posterior fetal position during the first stage of labour: a randomised controlled trial. BJOG. 2016 Dec;123(13):2199-2207. doi: 10.1111/1471-0528.13855. Epub 2016 Jan 24. PMID 26806596
- [Background] Choi SK, Park YG, Lee da H, Ko HS, Park IY, Shin JC. Sonographic assessment of fetal occiput position during labor for the prediction of labor dystocia and perinatal outcomes. J Matern Fetal Neonatal Med. 2016 Dec;29(24):3988-92. doi: 10.3109/14767058.2016.1152250. Epub 2016 Mar 7. PMID 26948718
- [Background] Khan KS. Optimal fetal positioning: a theory in tatters-time to rewrite textbooks. BJOG. 2016 Dec;123(13):2207. doi: 10.1111/1471-0528.13872. Epub 2016 Jan 25. No abstract available. PMID 26810973